CLINICAL TRIAL: NCT01083654
Title: Menominee Smoking Cessation Clinical Trial
Brief Title: Menominee Stop Tobacco Abuse Renew Tradition Study
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Wisconsin, Milwaukee (Other); Menominee Indian Tribe of Wisconsin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2009-0194
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Smoking
Keywords: Smoking; Smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treatment Counseling (Active Comparator): Standard Treatment (ST) will consist of 12 weeks of open-label varenicline and smoking cessation counseling consisting of four sessions: one in-person pre-quit counseling session during Study Visit 2, counseling during a phone call on the day after the quit day, and two additional in-person counseling sessions at Study Visits 3 and 4 (one week and three weeks after the quit day, respectively).
  Interventions: Behavioral: Standard Treatment Counseling
- Culturally-Tailored Treatment (Experimental): The Culturally-Tailored Treatment will consist of 12 weeks of open-label varenicline and culturally-tailored (for American Indians) smoking cessation counseling consisting of four sessions: one in-person pre-quit counseling session during Study Visit 2, counseling during a phone call on the day after the quit day, and two additional in-person counseling sessions at Study Visits 3 and 4 (one week and three weeks after the quit day, respectively).
  Interventions: Behavioral: Culturally-Tailored Treatment

INTERVENTIONS:
Behavioral: Standard Treatment Counseling — Standard Treatment Counseling will be based on recommendations in the 2008 U.S. Public Health Service Guideline (Treating Use and Dependence) including topics on preparing to quit, nicotine addiction, coping with stressors and challenging situations, coping with withdrawal symptoms, seeking support, and relapse prevention. Counseling will be delivered in an accessible, personalized manner by Ms. Fossum (an enrolled member of the Menominee Tribe) but no American Indian culturally-appropriate treatment elements will be incorporated into the counseling. In other words, the counseling in the Standard Treatment will be similar to the kind of evidence-based counseling offered to other smokers regardless of race or ethnicity.
  Arms: Standard Treatment Counseling
Behavioral: Culturally-Tailored Treatment — The Culturally-Tailored Treatment consists of the Standard Treatment Counseling plus culturally-appropriate treatment elements including: discussion of the long history of sacred/traditional use of tobacco (honoring and respecting native traditions) and how it differs from use of commercial tobacco use (harming health); custom booklet on smoking and smoking cessation tailored for Menominee and other American Indian smokers; and participants will be encouraged to make their own traditional tobacco pouch (symbol of long life)
  Arms: Culturally-Tailored Treatment

SUMMARY:
The purpose of this community-based study is to evaluate the effectiveness of a culturally-tailored smoking cessation treatment for American Indian (AI) smokers as compared to standard evidence-based cessation treatment (not culturally-tailored).

DETAILED DESCRIPTION:
Smoking is the leading preventable cause of illness and death. American Indians (AIs) have the highest rate of smoking but very little research has addressed how to help AIs quit smoking. AIs also suffer health disparities related to the addictive use of commercial tobacco. Many AIs also use natural tobacco for ceremonial purposes in addition to using commercial tobacco in an addictive manner. This study will add important new knowledge about how best to help AI smokers quit smoking (addictive use of commercial tobacco) and this is expected to help reduce the prevalence of smoking and smoking-related illness in AI communities. The "Menominee Smoking Cessation Clinical Trial" is a community-based study designed to evaluate a culturally-appropriate, evidence-based smoking cessation intervention for AI smokers. This project joins together collaborators at the University of Wisconsin Center for Tobacco Research and Intervention (UW-CTRI; PI Dr. Stevens Smith; smoking cessation expertise), the UW Carbone Comprehensive Cancer Center (UWCCC), the University of Wisconsin-Milwaukee (UWM; Dr. Leah Arndt; qualitative analysis expertise), and the Menominee Tribal Clinic (MTC; Wellness Director Mr. Mark Caskey; MTC Director Mr. Jerry Waukau, an enrolled member of the Menominee Tribe; and Ms. Jodi Fossum, an enrolled member of the Menominee Tribe) that serves Menominee and other AI patients. The study will randomize 150 AI smokers to two treatment conditions: (1) a standard evidence-based smoking cessation treatment condition (FDA-approved varenicline for 12 weeks + 4 counseling sessions), and, (2) a culturally-tailored smoking cessation treatment condition consisting of the standard treatment (FDA-approved varenicline for 12 weeks + 4 counseling sessions) plus culturally-appropriate treatment elements. Follow-up will be conducted at 3 and 6 months post-quit to assess smoking status and other study outcomes. We also plan to collect and analyze qualitative data (this aspect of the study will be led by Dr. Arndt) to learn more about the process and factors associated with cessation of commercial tobacco in American Indians including cultural factors.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age
2. must smoke cigarettes
3. eligible to receive health care services at the Menominee Tribal Clinic (i.e., must be an enrolled member of a federally-recognized American Indian Tribe)
4. primary care provider (M.D. or Nurse Practitioner) is at the Menominee Tribal Clinic
5. must be medically able and willing to take varenicline

Exclusion Criteria:

1. end-stage renal disease with hemodialysis
2. any prior suicide attempts
3. current or recent (past 12 months) suicidal ideation
4. currently pregnant or breastfeeding
5. unwilling to use appropriate methods of birth control while taking study medication and for 1 month after discontinuing study medication
6. primary care provider (PCP) determines that the individual should not take varenicline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stevens S. Smith, Ph.D., Principal Investigator — University of Wisconsin, Madison; Mark Caskey, B.S., R.N., Study Director — Menominee Tribal Clinic; Leah Arndt, Ph.D., Study Chair — University of Wisconsin, Milwaukee
Locations (1):
- Menominee Tribal Clinic, Keshena, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from February 22, 2010, to May 26, 2011 at the Menominee Tribal Clinic (MTC). The MTC Wellness Director or designee screened potential participants (adult American Indian smokers). Informed consent and HIPAA authorization were obtained at the Enrollment Visit.
Groups:
- Standard Treatment Counseling: Standard Treatment (ST) will consist of 12 weeks of open-label varenicline and smoking cessation counseling consisting of 4 sessions: one in-person pre-quit counseling session during Study Visit 2, counseling during a phone call on the day after the quit day, and two additional in-person counseling sessions at Study Visits 3 and 4 (one week and three weeks after the quit day, respectively).
  Standard Treatment Counseling: Standard Treatment Counseling will be based on recommendations in the 2008 U.S. Public Health Service Guideline (Treating Use and Dependence) including topics on preparing to quit, nicotine addiction, coping with stressors and challenging situations, coping with withdrawal symptoms, seeking support, and relapse prevention. Counseling will be delivered in an accessible, personalized manner by Ms. Fossum (an enrolled member of the Menominee Tribe) but no American Indian culturally-appropriate treatment elements will be incorporated into the counseling. In other w
- Culturally-Tailored Treatment: The Culturally-Tailored Treatment will consist of 12 weeks of open-label varenicline and culturally-tailored (for American Indians) smoking cessation counseling consisting of 4 sessions: one in-person pre-quit counseling session during Study Visit 2, counseling during a phone call on the day after the quit day, and two additional in-person counseling sessions at Study Visits 3 and 4 (one week and three weeks after the quit day, respectively).
  Culturally-Tailored Treatment: The Culturally-Tailored Treatment consists of the Standard Treatment Counseling plus culturally-appropriate treatment elements including: discussion of the long history of sacred/traditional use of tobacco (honoring and respecting native traditions) and how it differs from use of commercial tobacco use (harming health); custom booklet on smoking and smoking cessation tailored for Menominee and other American Indian smokers; and participants will be encouraged to make their own traditional tobacco pouch (symbol
Period: Overall Study
Arm/Group | Standard Treatment Counseling | Culturally-Tailored Treatment
Started | 53 | 50
Completed | 53 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adult American Indian smokers eligible for services at the Menominee Tribal Clinic.
Groups:
- Standard Treatment Counseling: Standard Treatment (ST) will consist of 12 weeks of open-label varenicline and smoking cessation counseling consisting of 4 sessions: one in-person pre-quit counseling session during Study Visit 2, counseling during a phone call on the day after the quit day, and two additional in-person counseling sessions at Study Visits 3 and 4 (one week and three weeks after the quit day, respectively).
  ST Counseling will be based on recommendations in the 2008 U.S. Public Health Service Guideline (Treating Use and Dependence) including topics on preparing to quit, nicotine addiction, coping with stressors and challenging situations, coping with withdrawal symptoms, seeking support, and relapse prevention. Counseling will be delivered in an accessible, personalized manner by an enrolled member of the Menominee Tribe but no American Indian culturally-appropriate treatment elements will be incorporated into the counseling.
- Culturally-Tailored Treatment: The Culturally-Tailored Treatment will consist of 12 weeks of open-label varenicline and culturally-tailored (for American Indians) smoking cessation counseling consisting of 4 sessions: one in-person pre-quit counseling session during Study Visit 2, counseling during a phone call on the day after the quit day, and two additional in-person counseling sessions at Study Visits 3 and 4 (one week and three weeks after the quit day, respectively).
  The Culturally-Tailored Treatment consists of the Standard Treatment Counseling plus culturally-appropriate treatment elements including: discussion of the long history of sacred/traditional use of tobacco (honoring and respecting native traditions) and how it differs from use of commercial tobacco use (harming health); custom booklet on smoking and smoking cessation tailored for Menominee and other American Indian smokers; and participants will be encouraged to make their own traditional tobacco pouch (symbol of long life)
- Total: Total of all reporting groups
Arm/Group | Standard Treatment Counseling | Culturally-Tailored Treatment | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (13.5) | 40.1 (12.7) | 39.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 19 | 20 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 53 | 50 | 103
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point-prevalence Smoking Abstinence
Description: Self-reported abstinence (versus smoking) during the past 7 days at the 6-month follow-up time-point, verified by exhaled breath carbon monoxide (CO) measurement (< 10 parts per million CO is indicative of no smoking).
Time Frame: 6 months
Measure: Number; unit: Number of abstinent participants
Groups:
- Culturally-Tailored Treatment: The Culturally-Tailored Treatment will consist of 12 weeks of open-label varenicline and culturally-tailored (for American Indians) smoking cessation counseling consisting of four sessions: one in-person pre-quit counseling session during Study Visit 2, counseling during a phone call on the day after the quit day, and two additional in-person counseling sessions at Study Visits 3 and 4 (one week and three weeks after the quit day, respectively).
  Culturally-Tailored Treatment: The Culturally-Tailored Treatment consists of the Standard Treatment Counseling plus culturally-appropriate treatment elements including: discussion of the long history of sacred/traditional use of tobacco (honoring and respecting native traditions) and how it differs from use of commercial tobacco use (harming health); custom booklet on smoking and smoking cessation tailored for Menominee and other American Indian smokers; and participants will be encouraged to make their own traditional tobacco pouch (symbol
Arm/Group | Standard Treatment Counseling | Culturally-Tailored Treatment
Number analyzed (Participants) | 53 | 50
Number of abstinent participants | 12 | 7
Statistical Analysis 1: Comparison: Standard Treatment Counseling vs Culturally-Tailored Treatment; Test type: Superiority or Other; p = .262, Regression, Logistic; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.20 to 1.55]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Medication adverse events were assessed during the 12 weeks of medication use.
Arm/Group | Standard Treatment Counseling | Culturally-Tailored Treatment
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 1/53 | 2/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment Counseling (N=53) | Culturally-Tailored Treatment (N=50)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Change in mood (Psychiatric disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes